CLINICAL TRIAL: NCT03028012
Title: Double-blind, Prospective Comparison of Medications Used in Trigger Point Injections - Ketorolac, Lidocaine, or Dexamethasone
Brief Title: TPI Medication Comparison - Ketorolac, Lidocaine, or Dexamethasone
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor enrollment.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Daniel Cushman, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 98370
Record Dates: First submitted 2017-01-14; First posted 2017-01-23 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Myofascial Pain
Keywords: Trigger Point Injections; steroid; nsaid
MeSH Terms: interventions — Ketorolac; Ketorolac Tromethamine; Lidocaine; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ketorolac (Experimental): Participants may be randomized to receive Ketorolac for their TPI.
  Interventions: Drug: Ketorolac
- Lidocaine (Experimental): Participants may be randomized to receive Lidocaine for their TPI.
  Interventions: Drug: Lidocaine
- Dexamethasone (Experimental): Participants may be randomized to receive Dexamethasone for their TPI.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Ketorolac — Participants may be randomized to receive Ketorolac for their TPI. This randomized study will compare the efficacy of the three substances used in TPIs.
  Other Names: Toradol
  Arms: Ketorolac
Drug: Lidocaine — Participants may be randomized to receive Lidocaine for their TPI. This randomized study will compare the efficacy of the three substances used in TPIs.
  Other Names: Xylocaine
  Arms: Lidocaine
Drug: Dexamethasone — Participants may be randomized to receive Dexamethasone for their TPI. This randomized study will compare the efficacy of the three substances used in TPIs.
  Other Names: Decadron
  Arms: Dexamethasone

SUMMARY:
Hypothesis

The main hypothesis of this study is that anti-inflammatory medications (ketorolac or dexamethasone) will provide longer-lasting and greater pain relief than just lidocaine in trigger point injections where a local twitch response is evoked at the time of the injection.

Purpose/Specific Aims

The primary objective of this study is to compare the efficacy of three substances used in TPIs with a LTR identified at the time of the injection: a CS (dexamethasone), a NSAID (ketorolac), or only a local anesthetic (lidocaine).

DETAILED DESCRIPTION:
Background

Trigger point injections (TPIs) are a commonly-performed procedures by physicians for the treatment of myofascial pain, specifically targeting myofascial trigger points (MTrPs). Commonly injected substances include local anesthetic, botulinum toxin, or corticosteroid (CS), though non-steroidal anti-inflammatory drugs (NSAIDs) and other substances have been reported. A Cochrane review found that intramuscular injection of local anesthetic demonstrated moderate evidence of benefit for mechanical neck disorders; no other treatment demonstrated greater benefit.

Great variation is seen in how TPIs are performed, however. The standard method was described by Simons and Travell, and is often cited. Hong et al. demonstrated that, similar to the technique described by Simons and Travell, obtaining a local twitch response (LTR) was the most important factor in producing pain relief. Further research by Shah et al., which demonstrated an inflammatory component to MTrPs, also showed a decrease in inflammatory cytokines following trigger point injections that obtained a LTR. Despite these findings, most studies do not use the LTR method in their TPI techniques.

Prior studies demonstrated that most patients obtain significant relief from TPI, but did not identify differences between injection of CS or other substances. However, none of these studies identified LTRs in their injection techniques.

As can be learned from a review of the published literature on muscular trigger points, the cause of this condition is unknown, and no single treatment approach has been established as a clearly accepted gold standard treatment. There is evidence, however, that there is an inflammatory component associated with trigger points and that obtaining a local twitch response is associated with a decrease in local inflammation at the site of a trigger point. The combination of injecting an anti-inflammatory medication and obtaining a local twitch response has never been studied. The purpose of this study is to examine the comparative effectiveness of injectable substances on patient outcome after a TPI with LTR identified, namely a CS (dexamethasone), a NSAID (ketorolac), or only a local anesthetic (lidocaine).

ELIGIBILITY:
Inclusion Criteria:

1. Men or women age 18 or over
2. At least one active trigger point

Exclusion Criteria:

1. Allergy or contraindication to any NSAID, CS, or local anesthetic
2. Receiving anticoagulant medication
3. History of bleeding disorder
4. Pregnant or breast feeding women
5. Gastrointestinal ulceration
6. Pre-existing renal disease
7. Pre-existing congestive heart failure
8. Diabetes mellitus
9. Prior myocardial infarction or stroke
10. Fibromyalgia

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Cushman, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hong CZ. Lidocaine injection versus dry needling to myofascial trigger point. The importance of the local twitch response. Am J Phys Med Rehabil. 1994 Jul-Aug;73(4):256-63. doi: 10.1097/00002060-199407000-00006. PMID 8043247
- [Background] Krishnan SK, Benzon HT, Siddiqui T, Canlas B. Pain on intramuscular injection of bupivacaine, ropivacaine, with and without dexamethasone. Reg Anesth Pain Med. 2000 Nov-Dec;25(6):615-9. doi: 10.1053/rapm.2000.8933. PMID 11097670
- [Background] Garvey TA, Marks MR, Wiesel SW. A prospective, randomized, double-blind evaluation of trigger-point injection therapy for low-back pain. Spine (Phila Pa 1976). 1989 Sep;14(9):962-4. doi: 10.1097/00007632-198909000-00008. PMID 2528826
- [Background] Frost FA, Jessen B, Siggaard-Andersen J. A control, double-blind comparison of mepivacaine injection versus saline injection for myofascial pain. Lancet. 1980 Mar 8;1(8167):499-500. doi: 10.1016/s0140-6736(80)92761-0. PMID 6102230
- [Background] McMillan AS, Nolan A, Kelly PJ. The efficacy of dry needling and procaine in the treatment of myofascial pain in the jaw muscles. J Orofac Pain. 1997 Fall;11(4):307-14. PMID 9656906
- [Background] Hameroff SR, Crago BR, Blitt CD, Womble J, Kanel J. Comparison of bupivacaine, etidocaine, and saline for trigger-point therapy. Anesth Analg. 1981 Oct;60(10):752-5. PMID 7027827
- [Background] Ay S, Evcik D, Tur BS. Comparison of injection methods in myofascial pain syndrome: a randomized controlled trial. Clin Rheumatol. 2010 Jan;29(1):19-23. doi: 10.1007/s10067-009-1307-8. Epub 2009 Oct 20. PMID 19838864
- [Background] Ga H, Koh HJ, Choi JH, Kim CH. Intramuscular and nerve root stimulation vs lidocaine injection to trigger points in myofascial pain syndrome. J Rehabil Med. 2007 May;39(5):374-8. doi: 10.2340/16501977-0058. PMID 17549328
- [Background] Misirlioglu TO, Akgun K, Palamar D, Erden MG, Erbilir T. Piriformis syndrome: comparison of the effectiveness of local anesthetic and corticosteroid injections: a double-blinded, randomized controlled study. Pain Physician. 2015 Mar-Apr;18(2):163-71. PMID 25794202
- [Background] Karadas O, Gul HL, Inan LE. Lidocaine injection of pericranial myofascial trigger points in the treatment of frequent episodic tension-type headache. J Headache Pain. 2013 May 22;14(1):44. doi: 10.1186/1129-2377-14-44. PMID 23698019
- [Background] Kamanli A, Kaya A, Ardicoglu O, Ozgocmen S, Zengin FO, Bayik Y. Comparison of lidocaine injection, botulinum toxin injection, and dry needling to trigger points in myofascial pain syndrome. Rheumatol Int. 2005 Oct;25(8):604-11. doi: 10.1007/s00296-004-0485-6. Epub 2004 Sep 15. PMID 15372199
- [Background] Wheeler AH, Goolkasian P, Gretz SS. A randomized, double-blind, prospective pilot study of botulinum toxin injection for refractory, unilateral, cervicothoracic, paraspinal, myofascial pain syndrome. Spine (Phila Pa 1976). 1998 Aug 1;23(15):1662-6; discussion 1667. doi: 10.1097/00007632-199808010-00009. PMID 9704373
- [Background] Cheshire WP, Abashian SW, Mann DJ. Botulinum toxin in the treatment of myofascial pain syndrome. Pain. 1994 Oct;59(1):65-69. doi: 10.1016/0304-3959(94)90048-5. PMID 7854804
- [Background] Benecke R, Heinze A, Reichel G, Hefter H, Gobel H; Dysport myofascial pain study group. Botulinum type A toxin complex for the relief of upper back myofascial pain syndrome: how do fixed-location injections compare with trigger point-focused injections? Pain Med. 2011 Nov;12(11):1607-14. doi: 10.1111/j.1526-4637.2011.01163.x. Epub 2011 Jun 21. PMID 21692970
- [Background] Gobel H, Heinze A, Reichel G, Hefter H, Benecke R; Dysport myofascial pain study group. Efficacy and safety of a single botulinum type A toxin complex treatment (Dysport) for the relief of upper back myofascial pain syndrome: results from a randomized double-blind placebo-controlled multicentre study. Pain. 2006 Nov;125(1-2):82-8. doi: 10.1016/j.pain.2006.05.001. Epub 2006 Jun 5. PMID 16750294
- [Background] Esenyel M, Caglar N, Aldemir T. Treatment of myofascial pain. Am J Phys Med Rehabil. 2000 Jan-Feb;79(1):48-52. doi: 10.1097/00002060-200001000-00011. PMID 10678603
- [Background] Tschopp KP, Gysin C. Local injection therapy in 107 patients with myofascial pain syndrome of the head and neck. ORL J Otorhinolaryngol Relat Spec. 1996 Nov-Dec;58(6):306-10. doi: 10.1159/000276860. PMID 8958538
- [Background] Cotchett MP, Landorf KB, Munteanu SE. Effectiveness of dry needling and injections of myofascial trigger points associated with plantar heel pain: a systematic review. J Foot Ankle Res. 2010 Sep 1;3:18. doi: 10.1186/1757-1146-3-18. PMID 20807448
- [Background] Desai MJ, Saini V, Saini S. Myofascial pain syndrome: a treatment review. Pain Ther. 2013 Jun;2(1):21-36. doi: 10.1007/s40122-013-0006-y. Epub 2013 Feb 12. PMID 25135034
- [Background] Soares A, Andriolo RB, Atallah AN, da Silva EM. Botulinum toxin for myofascial pain syndromes in adults. Cochrane Database Syst Rev. 2014 Jul 25;2014(7):CD007533. doi: 10.1002/14651858.CD007533.pub3. PMID 25062018
- [Background] Liu L, Huang QM, Liu QG, Ye G, Bo CZ, Chen MJ, Li P. Effectiveness of dry needling for myofascial trigger points associated with neck and shoulder pain: a systematic review and meta-analysis. Arch Phys Med Rehabil. 2015 May;96(5):944-55. doi: 10.1016/j.apmr.2014.12.015. Epub 2015 Jan 7. PMID 25576642
- [Background] Robbins MS, Kuruvilla D, Blumenfeld A, Charleston L 4th, Sorrell M, Robertson CE, Grosberg BM, Bender SD, Napchan U, Ashkenazi A; Peripheral Nerve Blocks and Other Interventional Procedures Special Interest Section of the American Headache Society. Trigger point injections for headache disorders: expert consensus methodology and narrative review. Headache. 2014 Oct;54(9):1441-59. doi: 10.1111/head.12442. Epub 2014 Aug 28. PMID 25168295
- [Background] Risser A, Donovan D, Heintzman J, Page T. NSAID prescribing precautions. Am Fam Physician. 2009 Dec 15;80(12):1371-8. PMID 20000300
- [Background] Tekin L, Akarsu S, Durmus O, Cakar E, Dincer U, Kiralp MZ. The effect of dry needling in the treatment of myofascial pain syndrome: a randomized double-blinded placebo-controlled trial. Clin Rheumatol. 2013 Mar;32(3):309-15. doi: 10.1007/s10067-012-2112-3. Epub 2012 Nov 9. PMID 23138883
- [Background] Kim DH, Yoon DM, Yoon KB. The effects of myofascial trigger point injections on nocturnal calf cramps. J Am Board Fam Med. 2015 Jan-Feb;28(1):21-7. doi: 10.3122/jabfm.2015.01.140151. PMID 25567819
- [Background] Gerber LH, Shah J, Rosenberger W, Armstrong K, Turo D, Otto P, Heimur J, Thaker N, Sikdar S. Dry Needling Alters Trigger Points in the Upper Trapezius Muscle and Reduces Pain in Subjects With Chronic Myofascial Pain. PM R. 2015 Jul;7(7):711-718. doi: 10.1016/j.pmrj.2015.01.020. Epub 2015 Feb 4. PMID 25661462
- [Background] Kietrys DM, Palombaro KM, Mannheimer JS. Dry needling for management of pain in the upper quarter and craniofacial region. Curr Pain Headache Rep. 2014;18(8):437. doi: 10.1007/s11916-014-0437-0. PMID 24912453
- [Background] Xie P, Qin B, Yang F, Yu T, Yu J, Wang J, Zheng H. Lidocaine Injection in the Intramuscular Innervation Zone Can Effectively Treat Chronic Neck Pain Caused by MTrPs in the Trapezius Muscle. Pain Physician. 2015 Sep-Oct;18(5):E815-26. PMID 26431135
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; CONSORT. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2012;10(1):28-55. doi: 10.1016/j.ijsu.2011.10.001. Epub 2011 Oct 12. PMID 22036893
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Qerama E, Fuglsang-Frederiksen A, Kasch H, Bach FW, Jensen TS. A double-blind, controlled study of botulinum toxin A in chronic myofascial pain. Neurology. 2006 Jul 25;67(2):241-5. doi: 10.1212/01.wnl.0000224731.06168.df. PMID 16864815
- [Background] Ojala T, Arokoski JP, Partanen J. The effect of small doses of botulinum toxin a on neck-shoulder myofascial pain syndrome: a double-blind, randomized, and controlled crossover trial. Clin J Pain. 2006 Jan;22(1):90-6. doi: 10.1097/01.ajp.0000151871.51406.c3. PMID 16340597
- [Background] De Andres J, Adsuara VM, Palmisani S, Villanueva V, Lopez-Alarcon MD. A double-blind, controlled, randomized trial to evaluate the efficacy of botulinum toxin for the treatment of lumbar myofascial pain in humans. Reg Anesth Pain Med. 2010 May-Jun;35(3):255-60. doi: 10.1097/AAP.0b013e3181d23241. PMID 20921836
- [Background] Kwanchuay P, Petchnumsin T, Yiemsiri P, Pasuk N, Srikanok W, Hathaiareerug C. Efficacy and Safety of Single Botulinum Toxin Type A (Botox(R)) Injection for Relief of Upper Trapezius Myofascial Trigger Point: A Randomized, Double-Blind, Placebo-Controlled Study. J Med Assoc Thai. 2015 Dec;98(12):1231-6. PMID 27004309
- [Background] Ashkenazi A, Young WB. The effects of greater occipital nerve block and trigger point injection on brush allodynia and pain in migraine. Headache. 2005 Apr;45(4):350-4. doi: 10.1111/j.1526-4610.2005.05073.x. PMID 15836572
- [Background] Frost A. Diclofenac versus lidocaine as injection therapy in myofascial pain. Scand J Rheumatol. 1986;15(2):153-6. doi: 10.3109/03009748609102082. PMID 3749828
- [Background] Shirokov VA, Potaturko AV, Zakharov IaIu. [Safety and efficacy of movalis injected into trigger points in lumbago-ischialgia syndrome]. Zh Nevrol Psikhiatr Im S S Korsakova. 2008;108(9):41-4. Russian. PMID 18833170
- [Background] Sternfeld M, Finkelstein Y, Hai E, Hod I. Tension headache treated by anti-inflammatory drug injected into GB 20 acupuncture point. Am J Chin Med. 1986;14(3-4):171-4. doi: 10.1142/S0192415X86000272. PMID 3799535
- [Background] Choi JW, Lee CJ, Lee SM, Shin BS, Jun B, Sim WS. Effect of Hyaluronidase Addition to Lidocaine for Trigger Point Injection in Myofascial Pain Syndrome. Pain Pract. 2016 Nov;16(8):1019-1026. doi: 10.1111/papr.12362. Epub 2015 Oct 7. PMID 26443389
- [Background] Yamaguchi A, Ogino Y, Iwakoshi C, Karasawa K, Ohki M. [Trigger point therapy for myofascial pain in cancer patients (second report) analysis results of special use-results surveillance by neovitacain(R) injection]. Gan To Kagaku Ryoho. 2012 Apr;39(4):605-11. Japanese. PMID 22504686
- [Background] Peloso P, Gross A, Haines T, Trinh K, Goldsmith CH, Burnie S; Cervical Overview Group. Medicinal and injection therapies for mechanical neck disorders. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD000319. doi: 10.1002/14651858.CD000319.pub4. PMID 17636629
- [Background] Shah JP, Phillips TM, Danoff JV, Gerber LH. An in vivo microanalytical technique for measuring the local biochemical milieu of human skeletal muscle. J Appl Physiol (1985). 2005 Nov;99(5):1977-84. doi: 10.1152/japplphysiol.00419.2005. Epub 2005 Jul 21. PMID 16037403
- [Background] Venancio Rde A, Alencar FG, Zamperini C. Different substances and dry-needling injections in patients with myofascial pain and headaches. Cranio. 2008 Apr;26(2):96-103. doi: 10.1179/crn.2008.014. PMID 18468269
- [Background] Simons DG, Travell JG, Simons LS. Travell & Simons' Myofascial Pain and Dysfunction: The Trigger Point Manual. Upper half of body. Vol. 1. Vol 1: Wolters Kluwer Health; 1999.
- [Background] Drewes AM, Andreasen A, Poulsen LH. Injection Therapy for Treatment of Chronic Myofascial Pain. J Musculoskelet Pain. 2010;1(3-4):289-294.

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketorolac: Participants may be randomized to receive Ketorolac for their TPI.
  Ketorolac: Participants may be randomized to receive 1mL of 1% lidocaine + 1mL of 30mg/mL Ketorolac for their TPI. Participants will be allowed to have subsequent injections, which is standard practice. They may receive up to four injections, spaced at least 1 week apart. This randomized study will compare the efficacy of the three substances used in TPIs.
- Lidocaine: Participants may be randomized to receive Lidocaine for their TPI.
  Lidocaine: Participants may be randomized to receive 2mL of 1% Lidocaine for their TPI. Participants will be allowed to have subsequent injections, which is standard practice39-43. They may receive up to four injections, spaced at least 1 week apart. This randomized study will compare the efficacy of the three substances used in TPIs.
- Dexamethasone: Participants may be randomized to receive Dexamethasone for their TPI.
  Dexamethasone: Participants may be randomized to receive 1mL of 1% lidocaine+1mL of 4mg/mL
  Dexamethasone for their TPI. Participants will be allowed to have subsequent injections, which is standard practice39-43. They may receive up to four injections, spaced at least 1 week apart. This randomized study will compare the efficacy of the three substances used in TPIs.
Period: Overall Study
Arm/Group | Ketorolac | Lidocaine | Dexamethasone
Started | 4 | 3 | 3
Completed | 2 | 0 | 0
Not Completed | 2 | 3 | 3
Not completed — Lost to Follow-up | 2 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketorolac | Lidocaine | Dexamethasone | Total
Number analyzed (Participants) | 4 | 3 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 2 | 8
  >=65 years | 1 | 0 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 54 [38 to 65] | 40 [33 to 54] | 47 [26 to 72] | 48 [26 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 8
  Male | 1 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasion | 4 | 3 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Responder Rate Greater Than 50% on the Numeric Rating Pain Scale (NRS) Improvement
Description: Participants in this study underwent TPIs by the following method. The needle was inserted into the trigger point with the goal of eliciting a local twitch responses(LTRs). When a LTR was obtained, 0.1mL of randomized drug was injected into that location within the muscle. This was repeated until LTRs disappeared, or 1.0mL had been injected, whichever came first. This was performed in a similar manner for all affected muscles, up to a maximum of 2mL. Participants self-report their brief pain inventory at each of their injections (up to four subsequent injections) based off of the standardized Numeric Rating pain Scale (NRS). The NRS is nationally recognized numeric scale from zero to ten, with zero being an example of no pain, one to three would demonstrate mild pain, four to six would be moderate pain, seven to nine would be severe pain and a ten would be the worst pain possible. Improvement in BPI was determined if their NRS score went down with each injection(s).
Time Frame: Pre-Post Injections Up to Three Months
Population: Participants in other ARM's did not complete survey
Measure: Count of Participants; unit: Participants
Arm/Group | Ketorolac | Lidocaine | Dexamethasone
Number analyzed (Participants) | 2 | 0 | 0
Participants | 1 | 0 | 0

2. Secondary Outcome: Numeric Rating Pain Scale (NRS) at Baseline and Three Months.
Description: TPI were treated with a needle inserted into the trigger point with the goal of eliciting a local twitch responses(LTRs). When a LTR was obtained, 0.1mL of randomized drug was injected into that location within the muscle. This was repeated until LTRs disappeared, or 1.0mL had been injected, whichever came first. Such was performed in a similar manner for all affected muscles, up to a maximum of 2mL. Participants self-report their brief pain inventory at each of their injections (up to four subsequent injections) based off of the standardized Numeric Rating pain Scale (NRS). The NRS is nationally recognized numeric scale from zero to ten, with zero being an example of no pain,one to three would demonstrate mild pain, four to six would be moderate pain, seven to nine would be severe pain and a ten would be the worst pain possible. Improvement in BPI was determined if their NRS score went down with each injection(s).
Time Frame: Pre-Injection and Three Month Post Injection(s)
Population: This study was terminated early due to low enrollment. Zero participants completed the Lidocaine and Dexamethasone arm.
Measure: Number; unit: score on a scale
Arm/Group | Ketorolac | Lidocaine | Dexamethasone
Number analyzed (Participants) | 2 | 0 | 0
score on a scale
  Participant Number 3 at Baseline | 8 |  |
  Participant Number 3 at 3 Months | 3 |  |
  Participant Number 8 at Baseline | 5 |  |
  Participant Number 8 at 3 Months | 3 |  |

3. Secondary Outcome: Brief Pain Inventory (BPI) - Modified
Description: The BPI was evaluated on a scale from 0-10. Zero would mean no interference and 10 would be calculated at complete interferences. We used a 7-point questionnaire about pain. All scores were calculated at baseline and three months.
Time Frame: Baseline and Three Months
Population: Participants in other ARM's did not complete surveys
Measure: Number; unit: score on a scale
Groups:
- Ketorolac: Participants may be randomized to receive Ketorolac for their TPI.
  Ketorolac: Participants may be randomized to receive 1mL of 1% lidocaine + 1mL of 30mg/mL Ketorolac for their TPI. Participants will be allowed to have subsequent injections, which is standard practice. Participants may receive up to four injections, spaced at least 1 week apart. This randomized study will compare the efficacy of the three substances used in TPIs.
Arm/Group | Ketorolac | Lidocaine | Dexamethasone
Number analyzed (Participants) | 2 | 0 | 0
score on a scale
  Participant Number #3 at Baseline | 8 |  |
  Participant Number #3 at 3 Months | 3 |  |
  Participant Number #8 at Baseline | 5 |  |
  Participant #8 at 3 Months | 3 |  |

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 3 month period.
Arm/Group | Ketorolac | Lidocaine | Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/3

LIMITATIONS AND CAVEATS:
Early termination of this study due to low subject enrollment, lack of participant follow-up to substantiated end of study measures. There was not enough reported data to provide statistically pertinent or relevant analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-04-05): https://cdn.clinicaltrials.gov/large-docs/12/NCT03028012/SAP_003.pdf
  • Study Protocol and Informed Consent Form (2017-04-05): https://cdn.clinicaltrials.gov/large-docs/12/NCT03028012/Prot_ICF_004.pdf